CLINICAL TRIAL: NCT03123783
Title: A Study to Evaluate the Safety and Efficacy of the CD40 Agonistic Antibody APX005M Administered in Combination With Nivolumab in Subjects With Non-small Cell Lung Cancer and Subjects With Metastatic Melanoma
Brief Title: CD40 Agonistic Antibody APX005M (Sotigalimab) in Combination With Nivolumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Apexigen America, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APX005M-002
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cancer; Non Small Cell Lung Cancer Metastatic; Metastatic Melanoma; Neoplasm of Lung; Melanoma
Keywords: CD40; Immunotherapy; Nivolumab; APX005M; PD-1
MeSH Terms: conditions — Neoplasms; Melanoma; Lung Neoplasms | interventions — sotigalimab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Phase 1b dose escalation with up to 4 sequential dose levels. Followed by Phase 2 dose expansion at Recommended Phase 2 Dose in 3 parallel disease cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1b escalation 0.03 mg/kg (Experimental): Non-small cell lung cancer (NSCLC) or metastatic melanoma
  APX005M 0.03 mg/kg and nivolumab 360 mg every 3 weeks
  Interventions: Drug: APX005M; Drug: Nivolumab
- Phase 1b escalation 0.1 mg/kg (Experimental): Non-small cell lung cancer (NSCLC) or metastatic melanoma
  APX005M 0.1 mg/kg and nivolumab 360 mg every 3 weeks
  Interventions: Drug: APX005M; Drug: Nivolumab
- Phase 1b escalation 0.3 mg/kg (Experimental): Non-small cell lung cancer (NSCLC) or metastatic melanoma
  APX005M 0.3 mg/kg and nivolumab 360 mg every 3 weeks
  Interventions: Drug: APX005M; Drug: Nivolumab
- Phase 2 expansion Cohort 1 (Experimental): Immunotherapy naïve, metastatic or locally advanced NSCLC
  APX005M 0.3 mg/kg and nivolumab 360 mg every 3 weeks
  Interventions: Drug: APX005M; Drug: Nivolumab
- Phase 2 expansion Cohort 2 (Experimental): Metastatic melanoma progressing during treatment with anti-PD-1/PD-L1 therapy
  APX005M 0.3 mg/kg and nivolumab 360 mg every 3 weeks
  Interventions: Drug: APX005M; Drug: Nivolumab
- Phase 2 expansion Cohort 3 (Experimental): Metastatic or locally advanced NSCLC progressing during treatment with anti-PD-1/PD-L1:
  * Group A: best response of progressive disease or with stable disease < 16 weeks
  * Group B: tumor response or with stable disease ≥ 16 weeks
  Interventions: Drug: APX005M; Drug: Nivolumab

INTERVENTIONS:
Drug: APX005M — APX005M is a CD40 agonistic monoclonal antibody
Drug: Nivolumab — Nivolumab is an immune checkpoint (PD-1) blocking antibody
  Other Names: Opdivo

SUMMARY:
This study is a Phase 1-2 open-label dose escalation study of the immuno-activating monoclonal antibody APX005M administered in combination with nivolumab to adult subjects with non-small cell lung cancer or metastatic melanoma. The Phase 1 portion is intended to establish the maximum tolerated dose and the recommended phase 2 dose of APX005M when administered in combination with nivolumab. The Phase 2 portion of the study will evaluate safety and efficacy of the combination.

DETAILED DESCRIPTION:
APX005M-002 is an open-label Phase 1-2 study and comprises a dose-escalation portion (Phase 1) followed by a Phase 2 tumor specific portion.

Eligible subjects with non-small cell lung cancer or metastatic melanoma will receive intravenous APX005M in combination with nivolumab until disease progression, unacceptable toxicity or death, whichever occurs first.

Study objectives include:

* Determine the maximum tolerated dose and the recommended phase 2 dose of APX005M when given in combination with nivolumab
* Evaluate safety of the APX005M and nivolumab combination
* Evaluate the objective response rate, duration of response and median PFS by RECIST 1.1 in subjects with non-small cell lung cancer or metastatic melanoma receiving APX005M in combination with nivolumab
* Determine the PK of APX005M

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, immunotherapy naïve or PD-1/PD-L1 pre-treated, metastatic or locally advanced non-small cell lung cancer not amenable to curative treatment. Subjects may be treatment naive or could have received one prior platinum based chemotherapy for non-small cell lung cancer and subjects with a documented activating mutation (e.g., EGFR, ALK, ROS) must also have received the appropriate therapy and progressed
* Histologically or cytologically confirmed unresectable or metastatic melanoma that progressed during treatment with an anti-PD-1/PD-L1 therapy and had confirmation of PD>=4 weeks later. Subjects with BRAF activating mutation could have also received a BRAF inhibitor and/or MEK inhibitor regimen prior to anti-PD-1/PD-L1 therapy.
* Measurable disease by RECIST 1.1
* ECOG performance status of 0 or 1
* Adequate bone marrow, liver and kidney function
* Negative pregnancy test for women of child bearing potential
* Agreement to use effective methods of contraception per the protocol requirements

Exclusion Criteria:

* Previous exposure to any immunomodulatory agents (e.g., anti- CD40, anti-PD-1/PD-L1, anti-CTLA-4, IDO inhibitors) except PD-1/PD-L1 targeting agents in the subsets of patients that must have previous treatment with anti-PD-1/PD-L1 therapy
* Second malignancy (solid or hematologic) within the past 3 years except locally curable cancers that have been apparently cured
* Active, known, clinically serious infections within the 14 days prior to first dose of investigational product
* Use of systemic corticosteroids or other systemic immunosuppressive drugs
* Active, known or suspected autoimmune disease
* History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis
* History of interstitial lung disease
* History of life-threatening toxicity related to prior anti-PD-1/PD-L1 treatment for subjects with metastatic melanoma or NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Pyxis Oncology, Inc
Locations (23):
- United States (13):
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - Yale University, New Haven, Connecticut
  - Hem-Onc Associates of the Treasure Coast, Port Saint Lucie, Florida
  - University of Maryland Marlene and Stewart Greenebaum Comprehensive Cancer Center (UMGCCC), Baltimore, Maryland
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - SUNY Upstate Medical Hospital, Syracuse, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Center, Rockledge, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
- Spain (10):
  - Hospital Quirón Dexeus, Barcelona
  - H. Vall d'Hebron, Barcelona
  - H. Clinic i Provincial, Barcelona
  - H. Insular de Gran Canaria, Las Palmas de Gran Canaria
  - H. Lucus Augusti, Lugo
  - H. Doce de Octubre, Madrid
  - H. HM Sanchinnarro, Madrid
  - H. de Málaga, Málaga
  - H. La Fe, Valencia
  - H. General de Valencia, Valencia de Alcántara

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Phase 1b dose-escalation portion of the study, a total of 10 participants were enrolled at 3 dose levels. Nine participants received at least one dose of both study drugs. 0.3 mg/kg was determined as the recommended phase 2 (RP2D) dose.
  Note: The 3 participants treated in DL3 of Phase 1b are at the RP2D and are also included in Phase 2 results. One participant was rolled over to Cohort 1 (Phase 2) and 2 participants were rolled over into Cohort 2 (Phase 2) to continue treatment.
Pre-assignment Details: For the phase 2 cohorts 1,2,3A,3B, a total of 133 participants were enrolled in 4 cohorts to receive APX005M at 0.3 mg/kg (RP2D) plus nivolumab at 360 mg IV. Three subjects who were treated at the RP2D in the Phase 1b dose-escalation portion of the study were included in Phase 2 of the relevant disease-specific cohort. The study enrollment was completed as planned and all primary and secondary outcome measures and adverse events were collected even though the study was ended by the sponsor.
Groups:
- DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b): Participants received 0.03mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg
- DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b): Participants received 0.1mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg
- DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b): Participants received 0.3 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg
- Cohort 1(Arm)/ inNSCLC (Phase 2); Cohort 2(Arm)/ PD1-MM (Phase 2) -; Cohort 3A(Arm)/ PD1-NSCLC (Phase 2); Cohort 3B(Arm)/ PD1-NSCLC (Phase 2): Participants received 0.3 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
Period: Phase 1b
Arm/Group | DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b) | DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b) | DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b) | Cohort 1(Arm)/ inNSCLC (Phase 2) | Cohort 2(Arm)/ PD1-MM (Phase 2) - | Cohort 3A(Arm)/ PD1-NSCLC (Phase 2) | Cohort 3B(Arm)/ PD1-NSCLC (Phase 2)
Started | 3 | 4 | 3 | 0 | 0 | 0 | 0
Participants in the Safety Population | 3 | 3 | 3 | 0 | 0 | 0 | 0
Participants in the Efficacy Population | 3 | 3 | 3 | 0 | 0 | 0 | 0
Completed (Participants completed Ph1b who did not receive RP2D did not roll over to Phase 2) | 3 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Removed from treatment prior to APX005M administration | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participants rolled over to Phase 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b) | DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b) | DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b) | Cohort 1(Arm)/ inNSCLC (Phase 2) | Cohort 2(Arm)/ PD1-MM (Phase 2) - | Cohort 3A(Arm)/ PD1-NSCLC (Phase 2) | Cohort 3B(Arm)/ PD1-NSCLC (Phase 2)
Started (Only 3 participants in Phase 1b rolled over to Phase 2 study) | 0 | 0 | 0 | 53 | 38 | 14 | 28
Phase 2 Participants in Safety Population | 0 | 0 | 0 | 53 | 38 | 14 | 28
Phase 2 Participants in the Efficacy (EE) Population | 0 | 0 | 0 | 48 | 33 | 12 | 25
Completed | 0 | 0 | 0 | 48 | 33 | 12 | 25
Not Completed | 0 | 0 | 0 | 5 | 5 | 2 | 3
Not completed — No post baseline tumor assesment on treatment period | 0 | 0 | 0 | 5 | 2 | 2 | 3
Not completed — Prior systemic therapy not allowed (1 patient did not complete post baseline tumor assessment) | 0 | 0 | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1b: immunotherapy naïve metastatic or locally advanced NSCLC (inNSCLC) or unresectable or metastatic melanoma (MM) Phase 2: Cohort 1/inNSCLC, Cohort 2/unresec or MM that progressed during treatment with anti-PD-1/PD-L1, Cohort 3/PD1-NSCLC metastatic or locally advanced NSCLC not amenable to curative treatment that progressed during prior treatment with anti-PD-1/PD-L1. Cohort 3A: best response of PD or with SD <16 wks, Cohort 3B includes PD1-NSCLC with tumor response or with SD ≥ 16 wks.
Groups:
- DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b): Participants received 0.03 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
- DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b): Participants received 0.1 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
- DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b); Cohort 1(Arm)/ inNSCLC (Phase 2); Cohort 2(Arm)/ PD1-MM (Phase 2); Cohort 3A(Arm)/ PD1-NSCLC (Phase 2); Cohort 3B(Arm)/ PD1-NSCLC (Phase 2): Participants received 0.3 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
- Total: Total of all reporting groups
Arm/Group | DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b) | DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b) | DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b) | Cohort 1(Arm)/ inNSCLC (Phase 2) | Cohort 2(Arm)/ PD1-MM (Phase 2) | Cohort 3A(Arm)/ PD1-NSCLC (Phase 2) | Cohort 3B(Arm)/ PD1-NSCLC (Phase 2) | Total
Number analyzed (Participants) | 3 | 4 | 3 | 52 | 36 | 14 | 28 | 140
Age, Categorical [Count of Participants; unit: Participants] — Population: The participants were enrolled into multiple Arms/Groups and are reported in the Arm/Group they were originally assigned.
  Participants
    Phase 1b Age, Categorical: number analyzed (Participants) | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 10
    Phase 1b Age, Categorical: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1b Age, Categorical: Between 18 and 65 years | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 6
    Phase 1b Age, Categorical: >=65 years | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 4
    Phase 2 Age, Categorical: number analyzed (Participants) | 0 | 0 | 0 | 52 | 36 | 14 | 28 | 130
    Phase 2 Age, Categorical: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 2 Age, Categorical: Between 18 and 65 years | 0 | 0 | 0 | 17 | 19 | 5 | 15 | 56
    Phase 2 Age, Categorical: >=65 years | 0 | 0 | 0 | 35 | 17 | 9 | 13 | 74
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The participants were enrolled into multiple Arms/Groups and are reported in the Arm/Group they were originally assigned
  Participants
    Phase 1b: number analyzed (Participants) | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 10
    Phase 1b: Female | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
    Phase 1b: Male | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 8
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 52 | 36 | 14 | 28 | 130
    Phase 2: Female | 0 | 0 | 0 | 21 | 15 | 5 | 9 | 50
    Phase 2: Male | 0 | 0 | 0 | 31 | 21 | 9 | 19 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The participants were enrolled into multiple Arms/Groups and are reported in the Arm/Group they were originally assigned
  Participants
    Phase 1b: number analyzed (Participants) | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 10
    Phase 1b: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1b: Not Hispanic or Latino | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 10
    Phase 1b: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 52 | 36 | 14 | 28 | 130
    Phase 2: Hispanic or Latino | 0 | 0 | 0 | 10 | 4 | 3 | 4 | 21
    Phase 2: Not Hispanic or Latino | 0 | 0 | 0 | 42 | 32 | 11 | 24 | 109
    Phase 2: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The participants were enrolled into multiple Arms/Groups and are reported in the Arm/Group they were originally assigned Population: The participants were enrolled into multiple Arms/Groups and are reported in the Arm/Group they were originally assigned
  Participants
    Phase 1b: number analyzed (Participants) | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 10
    Phase 1b: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1b: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1b: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1b: Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Phase 1b: White | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 9
    Phase 1b: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 1b: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 52 | 36 | 14 | 28 | 130
    Phase 2: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Phase 2: Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Phase 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 2: Black or African American | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 4
    Phase 2: White | 0 | 0 | 0 | 48 | 35 | 14 | 27 | 124
    Phase 2: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Phase 2: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 34 | 20 | 6 | 6 | 76
  Spain | 0 | 0 | 0 | 18 | 16 | 8 | 22 | 64
Weight [Mean (Full Range); unit: kg] — Population: The participants were enrolled into multiple Arms/Groups and are reported in the Arm/Group they were originally assigned
  kg
    Phase 1b: number analyzed (Participants) | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 10
    Phase 1b | 85.3 [67.4 to 112.5] | 84.33 [64.7 to 107.0] | 104.3 [93.4 to 118.4] |  |  |  |  | 90.63 [64.7 to 118.4]
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 52 | 36 | 14 | 28 | 130
    Phase 2 |  |  |  | 76.53 [50.26 to 106.59] | 80.15 [34.06 to 171.10] | 74.42 [55.00 to 95.60] | 71.80 [48.80 to 129.30] | 76.29 [34.06 to 171.10]
ECOG Performance Status [Count of Participants; unit: Participants] — Grade 0 - Normal activity, fully active, able to carry on all pre-disease performance without restriction Grade 1 - Symptoms, but fully ambulatory, restricted in physically strenuous but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work)
  Grade 0 is better than Grade 1. Population: The participants were enrolled into multiple Arms/Groups and are reported in the Arm/Group they were originally assigned
  Participants
    Phase 1b: number analyzed (Participants) | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 10
    Phase 1b: ECOG Score 0 | 1 | 1 | 3 |  |  |  |  | 5
    Phase 1b: ECOG Score 1 | 2 | 3 | 0 |  |  |  |  | 5
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 52 | 36 | 14 | 28 | 130
    Phase 2: ECOG Score 0 | 0 | 0 | 0 | 13 | 28 | 7 | 8 | 56
    Phase 2: ECOG Score 1 | 0 | 0 | 0 | 39 | 8 | 7 | 20 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-limiting Toxicities (DLTs)
Description: All toxicities were graded according to the NCI-CTCAE version 4.03. DLT was defined as any of the following events attributed to APX005M and nivolumab combination:
  * Grade 4 hematologic toxicity lasting ≥ 7 days (except asymptomatic lymphopenia)
  * Grade 3 or 4 neutropenia with a single temperature of >38.3◦ C (101◦ F) or a sustained temperature of ≥38◦ C (100.4◦ F) for more than one hour
  * Grade 4 thrombocytopenia or Grade ≥3 thrombocytopenia with signs or symptoms of bleeding or requiring platelet transfusion
  * Grade 4 non-hematologic toxicity
  * Grade 3 non-hematologic toxicity lasting >3 days despite optimal supportive care
  * Any Grade ≥ 3 non-hematologic laboratory value if: medical intervention is required to treat the subject, abnormality leads to hospitalization, or abnormality persists for >1 week
  * Failure to recover from a treatment-related AE to baseline or ≤ Grade 1 within 12 weeks of last dose of investigational product
  * Grade 5 toxicity.
Time Frame: Up to 21 days following first dose of APX005M and nivolumab
Population: All participants in the safety population who received at least 1 dose of study drug in the escalation cohorts (APX005M 0.03 mg/kg + nivolumab; APX005M 0.1 mg/kg + nivolumab; APX005M 0.3 mg/kg + nivolumab)
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b Escalation: Participants received intravenous infusions of APX005M starting at DL 0.03, .1 or .3 mg/kg administered every 21 days in combination with nivolumab 360 mg IV
Arm/Group | Phase 1b Escalation
Number analyzed (Participants) | 9
Participants | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of APX005M + Nivolumab (Phase 1b)
Description: Establish the MTD dose of APX005M combined with 360 mg of nivolumab for which for which < 33% of DLT- evaluable participants experience a DLT. In Phase 1b, the RP2D was based on the overall safety and tolerability of the combination of APX005M and nivolumab by testing increasing doses up to 0.3 mg/kg APX005M + nivolumab.
Time Frame: Up to 21 days following first dose of APX005M and nivolumab
Population: as for outcome 1
Measure: Number; unit: mg/kg
Arm/Group | Phase 1b Escalation
Number analyzed (Participants) | 9
mg/kg | NA — The MTD was formally not reached.

3. Primary Outcome: Phase 2 Evaluate the Objective Response Rate (ORR) by RECIST 1.1 and iRECIST in Each Cohort / Group
Description: ORR defined as the rate of patients who show as best overall response; either a complete response (CR) or a partial response (PR). The ORR can be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. using computed tomography (CT) scans/magnetic resonance imaging (MRI). Per RECIST v1.1, for target lesions and assessed by imaging: Complete Response, (CR), Disappearance of all target lesions and nontarget (NT) lesions; Partial Response (PR), >30% decrease in the sum of the longest diameter of target lesions and no PD in NT lesions or new lesions; Objective Response Rate (ORR)=CR + PR.
Time Frame: From start of the treatment (Day 1) until disease progression, withdrawal of consent, death, initiation of any anticancer therapy, lost to follow-up, or termination by the Sponsor, whichever comes first (for Phase 2: maximum up to 27 months)
Population: Cohort 1: immunotherapy naïve metastatic or locally advanced NSCLC, Cohort 2: unresectable or metastatic melanoma that progressed during treatment with anti-PD-1/PD-L1 therapy and had confirmation of PD ≥4 weeks, Cohort 3: PD1-NSCLC metastatic or locally advanced NSCLC not amenable to curative treatment that progressed during prior treatment with anti-PD-1/PD-L1 therapy. Cohort 3A: best response of PD or with SD <16 weeks, Cohort 3B includes PD1-NSCLC with tumor response or with SD ≥ 16 weeks
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 1 (Arm)/inNSCLC (Phase 2); Cohort 2(Arm)/PD1-MM (Phase 2); Cohort 3A(Arm)/PD1-NSCLC (Phase 2); Cohort 3B(Arm)/PD1-NSCLC (Phase 2): Participants received 0.3 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
Arm/Group | Cohort 1 (Arm)/inNSCLC (Phase 2) | Cohort 2(Arm)/PD1-MM (Phase 2) | Cohort 3A(Arm)/PD1-NSCLC (Phase 2) | Cohort 3B(Arm)/PD1-NSCLC (Phase 2)
Number analyzed (Participants) | 48 | 33 | 12 | 25
Percentage of participants | 16.67 [8.57 to 28.07] | 15.15 [6.17 to 29.25] | 0.00 [0.00 to 22.09] | 0.00 [0.00 to 11.29]

4. Secondary Outcome: Safety of the APX005M and Nivolumab Combination (Phase 2)
Description: Number of participants with TEAEs are reported.
Time Frame: Day 1 up to 30 days (or 100 days for SAEs and AEs with potential immunologic etiology) following the after the last dose of APX005M and/or nivolumab (from start of treatment up to 27 months)
Population: Any Adverse Event a participant has with two or more events in that category is counted only once
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Arm)/inNSCLC (Phase 2) | Cohort 2(Arm)/PD1-MM (Phase 2) | Cohort 3A(Arm)/PD1-NSCLC (Phase 2) | Cohort 3B(Arm)/PD1-NSCLC (Phase 2)
Number analyzed (Participants) | 53 | 38 | 14 | 28
Participants | 52 | 36 | 14 | 28

5. Secondary Outcome: Duration of Response (DOR) as Per RECIST 1.1(Phase 2)
Description: Duration of Response is defined as the time from the first evidence of confirmed partial response (PR) or better by Per RECIST v1.1 to disease progression or death due to any cause; in subjects alive without progressive disease (PD), DOR was censored on the date of the last tumor assessment. PD is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Maximum up to 25 months
Population: Cohort 1: immunotherapy naïve metastatic or locally advanced NSCLC, Cohort 2: unresectable or metastatic melanoma that progressed during treatment with anti-PD-1/PD-L1 therapy and had confirmation of PD ≥4 week. Cohort 3A/PD1-NSCLC and Cohort 3B/PD1 NSCLC had no objective response and therefore DOR could not be assessed.
Measure: Median (Full Range); unit: Months
Groups:
- Cohort 1(Arm)/inNSCLC (Phase 2); Cohort 2(Arm)/PD1-MM (Phase 2): Participants received 0.3 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
Arm/Group | Cohort 1(Arm)/inNSCLC (Phase 2) | Cohort 2(Arm)/PD1-MM (Phase 2)
Number analyzed (Participants) | 8 | 5
Months | NA [3.9 to 21.4] — NA because median duration of response not reached. | NA [4.2 to 24.7] — NA because median duration of response not reached. 4/5 participants had ongoing responses at the time of study closure.

6. Secondary Outcome: Median Progression-free Survival (PFS) (Phase 2)
Description: Progression-free Survival (PFS) in each cohort, measured from first dose to the earlier of PD (by RECIST 1.1) or death due to any cause, whichever occurs first.
Time Frame: From start of treatment (Day 1) up to 27 months
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1(Arm)/inNSCLC (Phase 2) | Cohort 2(Arm)/PD1-MM (Phase 2) | Cohort 3A(Arm)/PD1-NSCLC (Phase 2) | Cohort 3B(Arm)/PD1-NSCLC (Phase 2)
Number analyzed (Participants) | 48 | 33 | 12 | 25
Months | 4.11 [3.45 to 5.52] | 1.97 [1.87 to 3.61] | 3.43 [2.00 to 3.88] | 3.65 [1.84 to 3.81]

7. Secondary Outcome: 6-month PFS Rate (Phase 2)
Description: PFS rate in each cohort, measured from first dose to the earlier of PD (by RECIST 1.1) or death due to any cause, whichever occurs first.
Time Frame: * Outcome Measure Time Frame From start of treatment (Day 1) to 6 months
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1(Arm)/inNSCLC (Phase 2) | Cohort 2(Arm)/PD1-MM (Phase 2) | Cohort 3A(Arm)/PD1-NSCLC (Phase 2) | Cohort 3B(Arm)/PD1-NSCLC (Phase 2)
Number analyzed (Participants) | 48 | 33 | 12 | 25
Percentage of participants | 33.10 [20.10 to 46.68] | 21.21 [9.35 to 36.25] | 25.00 [6.01 to 50.48] | 12.92 [3.27 to 29.41]

ADVERSE EVENTS:
Time Frame: Day 1 through 30 days (or 100 days for SAEs and AEs with potential immunologic etiology) after the last dose of study drug (up to 27 months)
Description: An AE considered "serious" (SAE) if, in the view of either the Investigator or sponsor, it results in any of the following outcomes:
  * Death
  * A life-threatening AE
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital anomaly/birth defect
Groups:
- DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b Escalation): Participants received 0.03 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
- DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b Escalation): Participants received 0.1 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
- DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b Escalation): Participants received 0.3 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
  Note: One participant was rolled over to Cohort 1 (Phase 2) and 2 participants were rolled over into Cohort 2 (Phase 2).
- Cohort 1(Arm)/ inNSCLC (Phase 2) - Includes Data From 1 Participant From DL3; Cohort 2(Arm)/ PD1-MM (Phase 2) - Includes Data From 2 Participants From DL3; Cohort 3A(Arm)/ PD1-NSCLC (Phase 2); Cohort 3B(Arm)/ PD1-NSCLC (Phase 2): Participants received 0.3 mg/kg of APX005M administered every 21 days in combination with nivolumab 360 mg IV
Arm/Group | DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b Escalation) | DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b Escalation) | DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b Escalation) | Cohort 1(Arm)/ inNSCLC (Phase 2) - Includes Data From 1 Participant From DL3 | Cohort 2(Arm)/ PD1-MM (Phase 2) - Includes Data From 2 Participants From DL3 | Cohort 3A(Arm)/ PD1-NSCLC (Phase 2) | Cohort 3B(Arm)/ PD1-NSCLC (Phase 2)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 18/53 | 4/38 | 4/14 | 9/28
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 25/53 | 6/38 | 6/14 | 13/28
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 52/53 | 36/38 | 14/14 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b Escalation) (N=3) | DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b Escalation) (N=3) | DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b Escalation) (N=3) | Cohort 1(Arm)/ inNSCLC (Phase 2) - Includes Data From 1 Participant From DL3 (N=53) | Cohort 2(Arm)/ PD1-MM (Phase 2) - Includes Data From 2 Participants From DL3 (N=38) | Cohort 3A(Arm)/ PD1-NSCLC (Phase 2) (N=14) | Cohort 3B(Arm)/ PD1-NSCLC (Phase 2) (N=28)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infuenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL1 - APX005M 0.03 mg/kg + Nivolumab (Phase 1b Escalation) (N=3) | DL2 - APX005M 0.1 mg/kg + Nivolumab (Phase 1b Escalation) (N=3) | DL3 - APX005M 0.3 mg/kg + Nivolumab (Phase 1b Escalation) (N=3) | Cohort 1(Arm)/ inNSCLC (Phase 2) - Includes Data From 1 Participant From DL3 (N=53) | Cohort 2(Arm)/ PD1-MM (Phase 2) - Includes Data From 2 Participants From DL3 (N=38) | Cohort 3A(Arm)/ PD1-NSCLC (Phase 2) (N=14) | Cohort 3B(Arm)/ PD1-NSCLC (Phase 2) (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 13 (31) | 4 (8) | 0 (0) | 6 (10)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 7 (7) | 2 (2) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (7) | 2 (2) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 10 (15) | 5 (5) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 12 (37) | 6 (8) | 2 (8) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (7) | 3 (5) | 24 (54) | 18 (22) | 7 (13) | 8 (13)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (4) | 18 (46) | 10 (19) | 2 (3) | 5 (8)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 6 (10) | 4 (6) | 12 (17)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (8)
Chills (General disorders) | 0 (0) | 2 (3) | 3 (5) | 30 (65) | 19 (51) | 5 (14) | 13 (24)
Fatigue (General disorders) | 3 (4) | 2 (8) | 0 (0) | 18 (41) | 15 (36) | 5 (12) | 4 (4)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (4) | 0 (0) | 4 (7) | 3 (3) | 3 (3) | 2 (2)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 2 (4) | 28 (56) | 26 (57) | 7 (34) | 12 (24)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 3 (4) | 2 (2) | 3 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 11 (33) | 11 (19) | 4 (6) | 8 (34)
Blood alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 9 (34) | 7 (12) | 1 (1) | 3 (5)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 3 (5) | 0 (0) | 1 (4)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 1 (5) | 1 (2) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (19) | 7 (18) | 4 (10) | 5 (15)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (7) | 0 (0) | 3 (3)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (10) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 14 (21) | 0 (0) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (9) | 1 (2) | 14 (15) | 4 (4) | 4 (5) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (10) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (5) | 12 (23) | 6 (16) | 3 (3) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 8 (11) | 4 (6) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 4 (4) | 6 (10) | 1 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (6) | 0 (0) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 8 (13) | 8 (20) | 2 (4) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 13 (14) | 1 (1) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 13 (16) | 3 (4) | 3 (3) | 10 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 21 (30) | 3 (3) | 6 (8) | 8 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 16 (34) | 13 (15) | 4 (7) | 4 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (3) | 9 (13) | 10 (13) | 1 (3) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (9) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 3 (3) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (16) | 2 (2) | 0 (0) | 3 (5)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 10 (16) | 4 (5) | 1 (1) | 3 (4)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (4) | 1 (2) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (5) | 0 (0) | 12 (23) | 9 (16) | 4 (5) | 8 (17)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decrease (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monocyte count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal exudates (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Pharygitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood cortisol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ostenonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruitus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
In the AE section, DL3 participant data had no DLTs; AE data collected from DL3 was also added to Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT03123783/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03123783/SAP_001.pdf